CLINICAL TRIAL: NCT04140461
Title: Antifungal Treatment of Cryptococcal Meningitis
Brief Title: AmB Dose for Cryptococcal Meningitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Jun Chen, Assistant of the department, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMBDOSE
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Cryptococcal Meningitis; HIV Infections
Keywords: HIV infection; Cryptococcal Meningitis; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections | interventions — Amphotericin B; Antiretroviral Therapy, Highly Active; Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial (Experimental): Amphotericin B 0.5 mg/kg IVGTT QD + Flucytosine 100mg/kg PO QD for 4 weeks
  Interventions: Drug: Amphotericin B; Drug: Flucytosine
- Control (Active Comparator): Amphotericin B 0.7 mg/kg IVGTT QD + Flucytosine 100mg/kg PO QD for 2 weeks
  Interventions: Drug: Amphotericin B; Drug: Flucytosine

INTERVENTIONS:
Drug: Amphotericin B — The trial group and the control group received AmB 0.5mg/kg for 4 weeks and 0.7mg/kg for 2 weeks respectively.
  Other Names: Antiretroviral therapy
Drug: Flucytosine — The trial group and the control group received 100mg/kg for 4 weeks and for 2 weeks respectively.

SUMMARY:
Cryptococcal meningitis (CM) is one of the leading opportunistic infections and one of the most common causes of death in AIDS patients.

Amphotericin B (AmB) is the corner stone in CM treatment. The effect of AmB was dose-dependent. Recent retrospective study indicated that longer duration rather than higher dose of AmB is necessary to reduce the mortality of CM. We aimed to explore the efficacy and safety of small dose but longer duration of AmB for the treatment of HIV-associated CM.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Naive to antiretroviral therapy
* Cryptococcal antigen, smear or culture positive in cerebrospinal fluid
* Agree to participate the study

Exclusion Criteria:

* Having receiving antifungal treatment for ≥3 days
* ALT or AST > 5* upper limit of detection (ULD), or neutrophil< 0.5*10E9 cells/L, or hemoglobin < 90g/L or platelet <50*10E9/L or serum creatinine > ULD
* Pregnancy or breastfeeding
* Concomitant medications that are contraindicated with any research drug
* Any other contraindications for using amphotericin B or 5FC
* Inability to follow-up as accessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-02 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects died at weeks 48 | 48 weeks after randomization
  Mortality in intent to treat population

SECONDARY OUTCOMES:
Number of subjects with CSF culture positive for Cryptococcus at weeks 2 | 2 weeks after randomization
  Antifungal Activity
Number of subjects with disability at weeks 48 | 48 weeks after randomization
  Disability rate in intent to treat population

OTHER OUTCOMES:
Treatment-Emergent Adverse Events | 12 weeks after randomization
  All the adverse events occurred after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China